CLINICAL TRIAL: NCT06604572
Title: Clinical Study of Transabdominal Preperitoneal Approach Versus Open Tension-free Hernia Repair for the Treatment of Recurrent Inguinal Hernia
Brief Title: TAPP and Open Repair for Recurrent Inguinal Hernia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Weiming Li, director, The Second Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PJ-2022-85
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Recurrent Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transabdominal preperitoneal approach surgery group (Experimental): The enrolled patients were treated with Transabdominal preperitoneal approach
  Interventions: Procedure: Transabdominal preperitoneal approach
- Open tension-free hernia repair group (Other): The enrolled patients were treated with open tension-free hernia repair
  Interventions: Procedure: Transabdominal preperitoneal approach

INTERVENTIONS:
Procedure: Transabdominal preperitoneal approach — The enrolled patients underwent either open tension-free hernia repair or Transabdominal preperitoneal approach
  Other Names: Open tension-free hernia repair

SUMMARY:
The objective of this study was to explore the clinical efficacy of transabdominal preperitoneal approach (TAPP) and open tension-free hernia repair in the treatment of recurrent inguinal hernia. This study aims to provide a basis for selecting the optimal treatment methods for recurrent hernias.

DETAILED DESCRIPTION:
The patients were randomly allocated to the TAPP group and the open tension-free repair group. We recorded the general situation, operation time, and intraoperative complications; postoperative visual analogue pain scale (VAS) scores at 24 and 48 h; and the incidence of complications such as seroma, chronic pain, inguinal numbness, foreign body sensation, and recurrence at 1 week, 1 month, 3 months, 6 months and 1 year after surgery. These indicators were compared between the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* the diagnosis of recurrent inguinal hernia made by ultrasound or computed tomography (CT) during the present visit
* ability to tolerate general anesthesia and local anesthesia surgery
* all patients and their families agreed to participate in this study and sign relevant informed consent.

Exclusion Criteria:

* patch infection during the first surgery
* multiple (≥ 2) relapses
* inability to cooperate to complete follow-up after surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-28 (Estimated)

PRIMARY OUTCOMES:
Postoperation pain | 24 hours, 48 hours, three months after surgery
  Postoperative pain was monitored using the VAS pain scoring system (0-10 points) and recorded at 24 and 48 h. Patients with groin pain for more than 3 months were recorded during follow-up.

SECONDARY OUTCOMES:
Numbness and foreign body sensation | The mean follow-up time was 10 months after surgery
  The occurrence of groin numbness and foreign body sensation after operation was recorded
Operating time | During surgery
  Record the patient's operating time
Hemorrhage | During surgery
  The amount of surgical bleeding was recorded
Urinary retention | One week after surgery
  Urinary retention was observed and recorded after operation
Seroma | The mean follow-up time was 2 weeks after surgery
  The occurrence of postoperative seroma was observed and recorded
Recurrence | The mean follow-up time was 1 year after surgery
  The recurrence of patients after operation was observed and recorded
Fever | One week after surgery
  The postoperative fever was observed and recorded
Length of hospital stay | Within a week of surgery
  The patient's length of stay was recorded

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Li, doctor, Principal Investigator — The Second Affiliated Hospital of Kunming Medical University
Locations (1):
- Clinical study of recurrent inguinal hernia, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided